CLINICAL TRIAL: NCT02844114
Title: Clinical Study of Ganoderma Lucidum Spore Combined With Chemotherapy
Acronym: LCKY2015-21(x)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gao Yajie (Other)
Responsible Party: Sponsor-Investigator, Gao Yajie, Clinical Professor, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NationalHealthyFood G20090069
Record Dates: First submitted 2016-06-19; First posted 2016-07-26 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Ganoderma Lucidum Spore; Carcinoma, Non-Small-Cell Lung; Chemotherapy; Gemcitabine; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganoderma lucidum spore & Chemotherapy (Experimental): Ganoderma lucidum spore 1500mg tablet by mouth, every 8 hours for 7 days; Gemcitabine 1000mg intravenously on days 1 and 8 every 3 weeks(iv.over 30 minutes) or cisplatin 75mg intravenously on days 2 and 3 every 3 weeks (iv.15-30 minutes).
  Interventions: Drug: Ganoderma lucidum spore; Drug: Chemotherapy
- Placebo & Chemotherapy (Placebo Comparator): Placebo tablet by mouth, every 8 hours for 7 days; Gemcitabine 1000mg intravenously on days 1 and 8 every 3 weeks(iv.over 30 minutes) or cisplatin 75mg intravenously on days 2 and 3 every 3 weeks (iv.15-30 minutes).
  Interventions: Drug: Placebo; Drug: Chemotherapy

INTERVENTIONS:
Drug: Ganoderma lucidum spore — G 300mg, 5 tablets by mouth
  Other Names: G
  Arms: Ganoderma lucidum spore & Chemotherapy
Drug: Placebo — Sugar pill manufactured to mimic tramadol 1500mg tablet
  Other Names: P
  Arms: Placebo & Chemotherapy
Drug: Chemotherapy — iv.30 minutes
  Other Names: Gemcitabine, Cisplatin

SUMMARY:
This study evaluates the effect of the serum level of Superoxide Dismutase (SOD), Malondialdehyde (MDA), pro-inflammatory factors, stress hormones and Glutathione peroxidase (GSH-PX)in tumor patients with the treatment of Ganoderma lucidum spore based combination chemotherapy. Half of participants will receive Ganoderma lucidum spore and chemotherapy in combination, and the other half will receive a placebo and chemotherapy.

Study design: Phase 2. Experimental: Ganoderma lucidum spore & Chemotherapy; Placebo Comparator: Placebo & Chemotherapy.

Outcome Measure:

1. The life quality of participants was assessed with use of the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire at the initial diagnosis (baseline) and at 42 days after the treatment;
2. Investigators assessed Procedural mortality factor ligand 1(PD-L1)expression prospectively on tumour cells and tumour-infiltrating immune cells with the VENTANA PD-L1 immunohistochemistry assay;
3. National Cancer Institute Common Toxicity Criteria.

Statistical analysis: All experiment results were analyzed with Statistical Product and Service Solutions (SPSS) software (version 16.0). Data are presented as mean±standard deviation and analysed by one-way ANOVA. Semi-quantitative data were compared using the Kruskal- Wallis nonparametric analysis. The results were considered statistically significant at P<0.05.

DETAILED DESCRIPTION:
Ganoderma lucidum spore, as a natural substance is widely recognized and used in tumor patients for its nutritive value. The effect has proved that Ganoderma lucidum spore which has polysaccharide, triterpene compounds and the other trace elements, combined with chemotherapy can reduce toxicity and enhance efficacy in patients.

Ganoderma lucidum spore can reduce bone narrow depression, gastrointestinal mucosal damage and enhance the immunity. Previous studies have reported that Ganoderma lucidum spore have antivirus, antineoplastic, decreasing blood lipids, hypoglycemic and anti-hypoxic activities. The objective of this study is to observe the effect of Ganoderma lucidum spore based combination chemotherapy in treatment of patients. And then to detect the serum level of SOD, MDA, pro-inflammatory factors, stress hormones and GSH-PX.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed definitely by cytopathology examination and image methods.
* Eastern Cooperative Oncology Group (ECOG) score standard: 0-2.
* Survival time may last more than 3 months.
* Normal electrocardiogram changes.
* WBC≧4.0×10*9/L, PLT≧1.5×10*9/L, HB≧100.0g/L
* Have no cardiac disease, no myocardial infarction in past 6 months.

Exclusion Criteria:

* Receiving other effective treatments currently.
* Have diabetes or another chronic metabolic disorder (BIM <18 or >25).
* Serious pyogenic or chronic infections.
* Have hematologic disease or coagulation dysfunction.
* Unhealed serious cerebral disease or tumor, depression disorders, senile dementia or other mental diseases.
* Pregnant and lactation women, allergic constitution.
* Combined liver, kidney, blood system Primary serious diseases, mental patients.
* Within the past 4 weeks to participate in other clinical trials of patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The life quality of participants was assessed with use of the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire at the initial diagnosis (baseline) and at 42 days after the treatment. | 42 days

SECONDARY OUTCOMES:
Investigators assessed Procedural mortality factor ligand 1(PD-L1) expression prospectively on tumour cells and tumour-infiltrating immune cells with the VENTANA PD-L1 immunohistochemistry assay. | 42 days
  Investigators scored tumour cells expressing PD-L1 as a percentage of total tumour cells and tumour-infiltrating immune cells expressing PD-L1 as a percentage of tumour area, as previously described (tumour cells scored as percentage of PD-L1-expressing tumour cells)

OTHER OUTCOMES:
Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to National Cancer Institute Common Toxicity Criteria | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Yajie Gao, Professor, Study Chair — First Hospital of Dalian Medical University
Locations (1):
- First Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures within 6 months of study completion.